CLINICAL TRIAL: NCT02867423
Title: PHASE II STUDY : Hypofractionated Radiation by CyberKnife as a Mean of Radiation of the Tumor Site After Conventional Breast Radiation.
Brief Title: Hypofractionated Radiation by CyberKnife as a Mean of the Tumor Site's Radiation After Conventional Breast Radiation.
Acronym: CYBERBOOST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Antoine Lacassagne (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009/01 CYBERBOOST; 2010-A00284-35 (Other: AFSSAPS ID RCB)
Record Dates: First submitted 2016-08-11; First posted 2016-08-16 (Estimated); Last update posted 2025-09-30 (Actual); Status verified 2017-11

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A - CK boost radiation (Other): CK boost radiation
  Interventions: Device: CK Boost radiation

INTERVENTIONS:
Device: CK Boost radiation — single dose of 8 Grays is issued by the CK to the 6th week after conventional radiation

SUMMARY:
The CyberKnife (CK) has been developed recently. This is a linear accelerator carried by an industrial robot. It has, due to its tumor tracking capabilities and high accuracy, an interest in irradiation (boost) of tumor site after conventional irradiation. The radiation boost is currently issued by electrons, protons or brachytherapy. These techniques require several fractions and are associated with cutaneous toxicities and aesthetic problems. CK has an interest in reducing the number of fractions and a reduction of dose delivered to the skin.

CK has been used in a phase I protocol (CYBERNEO) with concomitant chemotherapy for inoperable breast tumors and has proven its effectiveness and safety of treatments.

The investigator is considering conducting a Phase II protocol to a single dose of 8 Grays issued by CK for boost to the tumor site after conventional breast irradiation.

The results, in terms of local control, will be evaluated on clinical monitoring.

ELIGIBILITY:
Inclusion Criteria:

1. unifocal breast cancer histologically proven
2. Age> 18 years old, in good general condition (ECOG 0-2)
3. No cons-indication for radiotherapy
4. Patient who underwent lumpectomy and axillary dissection or sentinel node technique.
5. carcinoma histology ductal or lobular carcinoma
6. surgical margins microscopically without residual disease (> 1 mm)
7. tumors classes T1 or T2, N0

Exclusion criteria

1. residual calcifications on X-ray examination
2. Inflammatory breast cancer, ductal (and / or in situ) and invasive lobular
3. multifocal breast Cancer
4. prior Breast radiotherapy
5. Patient who received chemotherapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2011-02; Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
EORTC score for erythema, telangiectasia, edema, pain | 2 months
  early skin toxicity evaluation by clinical examination (radiation oncology and dermatologist) using EORTC score for erythema, telangiectasia, edema, pain.

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Yves BONDIAU, md, Principal Investigator — Centre Antoine Lacassagne
Locations (1):
- Centre Antoine LACASSAGNE, Nice, France

IPD SHARING:
Plan to Share IPD: Undecided